CLINICAL TRIAL: NCT03584685
Title: The Impact of the Surgical Mask on the Relationship Between Patient and Family Nurse in Primary Care
Brief Title: Impact of the Surgical Mask on the Patient-nurse Relation in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: MASK
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-06

CONDITIONS: Satisfaction, Personal
MeSH Terms: conditions — Personal Satisfaction | interventions — Masks

STUDY DESIGN:
Intervention Model Description: All participants will initially be treated without the surgical mask. Then, half will be treated with the mask and the other half will be treated without the mask.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are blind as to whether they are in the control or experimental groups. The investigators and outcomes assessors are blind to which patients received the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Mask (Experimental): Use of the surgical mask in one routine wound treatment appointment.
  Interventions: Device: Mask
- Without Mask (Active Comparator): Routine wound treatment appointment without nurses wearing the surgical mask.
  Interventions: Procedure: Routine wound treatment

INTERVENTIONS:
Device: Mask — All participants will initially be treated without the mask. In the next appointment, half will be treated with the mask.
  Arms: With Mask
Procedure: Routine wound treatment — All participants will initially be treated for their wounds without the mask. In the next appointment, half will again be treated for their wounds without the mask.
  Arms: Without Mask

SUMMARY:
The goal of this study is to inspect the effect of nurses wearing the surgical mask on their patients' satisfaction with the relationship. All participants will initially be treated without the mask. Then, half will be treated with the mask and the other half will be treated without the mask.

DETAILED DESCRIPTION:
The use of the surgical mask has well-known benefits for both the patient and the professional regarding the control of infection contamination. However, its use is left to individual criteria, and is passed on from generation to generation of nurses through experiential, intuitive knowledge. Studies are necessary to support the use of the surgical mask.

Research indicates that wearing the mask affects perception of words, thus influencing patient-nurse communication. However, it might also affect the very nurse--patient relation. For example, it can convey the idea of personal distancing, which can either be appreciated by patients as dutiful professional care by the nurse, or viewed as a limit imposed on interpersonal communication and on the relationship.

This study inspects patient satisfaction about (1) interpersonal aspects and (2) professionalism in the patient-nurse relationship when the mask is used.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from chronic wounds
* Age: 18 years or older
* Know how to read and write in Portuguese
* Confirmed autopsychic and allopsychic orientation
* Maintain previous relation with the nurse of at least 18 months
* Need at least two consecutive treatments with the nurse

Exclusion Criteria:

* Failing to meet the above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
30-item questionnaire assessing patient satisfaction with the nurse-patient relation (the PSQ-III) | 1 day
  Self-reported patient satisfaction after one appointment with the nurse about interpersonal aspects of the patient-nurse relation (7 items), communication (5 items) and nurse's technical quality (10 items). Responses are given on a 1 to 5 Likert scale. Higher scores correspond to greater satisfaction.

SECONDARY OUTCOMES:
Sensation of time | 1 day
  1 question asked about how long patients and nurses felt that the appointment lasted

CONTACTS AND LOCATIONS:
Overall Officials: Irene P Carvalho, PhD, Principal Investigator — CINTESIS, Faculty of Medicine, University of Porto
Locations (1):
- CINTESIS - Faculty of Medicine of the University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No